CLINICAL TRIAL: NCT04346693
Title: An Open Randomized Study of Dalargin Efectiveness in Combination With Leitragin Drug for the Prevention and Treatment of Symptoms of Pulmonary Complications in Patients With Coronavirus Infection (SARS-COVID-19)
Brief Title: An Open Randomized Study of Dalargin Efectiveness in Combination With Leitragin Drug in Patients With Severe and Critical Manifestations of SARS-COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Burnasyan Federal Medical Biophysical Center (Other Government)
Responsible Party: Principal Investigator, Tatyana Astrelina, MD PhD, DSc (medicine), Head of Center for Biomedical Technologies State Research Center Burnasyan Federal Medical Biophysical Center FMBA of Russia, Burnasyan Federal Medical Biophysical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DAL-05-04-2020
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Acute Respiratory Tract Infection; Acute Respiratory Insufficiency; Pneumonia; Septic Shock; Hypoxemia
MeSH Terms: conditions — Pneumonia; Shock, Septic; Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Active Comparator): 80 patients with moderate and critical severity of the COVID19 with respiratory symptoms without Acute Respiratory Distress Syndrome (ADRS). Standard therapy is prescribed recommended by the Ministry of Health of the Russian Federation.
  Interventions: Procedure: Standard therapy recommended by the Ministry of Health of the Russian Federation.
- group 2 (Experimental): 80 patients with moderate to critical severity of the COVID19 with respiratory symptoms without Acute Respiratory Distress Syndrome (ADRS). A standard concomitant therapy will be given recommended by the Ministry of Health of the Russian Federation, with the additional intramuscular injection of the drug Dalargin (solution for intravenous and intramuscular doses of 1 mg once a day for 10 days).
  Interventions: Procedure: Standard therapy recommended by the Ministry of Health of the Russian Federation and Leitragin intramuscular injection
- group 3 (Experimental): 80 patients with moderate to critical severity of the COVID19 with respiratory symptoms without Acute Respiratory Distress Syndrome. A standard concomitant therapy will be given recommended by the Ministry of Health of the Russian Federation, with the additional inhalation of the drug Leitragin, at a dose of 10 mg daily once a day until the symptoms of pulmonary complications will be ceased.
  Interventions: Procedure: Standard therapy recommended by the Ministry of Health of the Russian Federation and Leitragin inhalation
- group 4 (Experimental): 80 patients with moderate to critical severity of the disease with respiratory symptoms without Acute Respiratory Distress Syndrome. A standard concomitant therapy will be given recommended by the Ministry of Health of the Russian Federation, with the additional intramuscular administration of the drug Dalargin (solution for intravenous and intramuscular doses of 1 mg once a day for 10 days) in conjunction with inhalation of the drug Leitragin, at a dose of 10 mg daily once a day until the symptoms of pulmonary complications will be ceased.
  Interventions: Procedure: Standard therapy recommended by the Ministry of Health of the Russian Federation and Leitragin intramuscular injection combined with Leitragin inhalation

INTERVENTIONS:
Procedure: Standard therapy recommended by the Ministry of Health of the Russian Federation. — Hydroxychloroquine + azithromycin + / - tocilizumab. Hydroxychloroquine intake is conducted according to the following schedule: 400 mg twice per day for 1-2 days of the treatment and 200 mg twice per day during six days of the treatment course.
  For the tocilizumab, 400 mg intravenously drip slowly (for at least 1 hour), with insufficient effect, administration is repeated the after 12 hours. Simultaneously no more than 800 mg of tocilizumab could be administered.
  For the azithromycin admission 500mg on day 1 is prescribed followed by 250mg per day, the next four days
  Arms: group 1
Procedure: Standard therapy recommended by the Ministry of Health of the Russian Federation and Leitragin intramuscular injection — Hydroxychloroquine + azithromycin + / - tocilizumab. Hydroxychloroquine intake is conducted according to the following schedule: 400 mg twice per day for 1-2 days of the treatment and 200 mg twice per day during six days of the treatment course.
  For the tocilizumab, 400 mg intravenously drip slowly (for at least 1 hour), with insufficient effect, administration is repeated the after 12 hours. Simultaneously no more than 800 mg of tocilizumab could be administered.
  For the azithromycin admission 500mg on day 1 is prescribed followed by 250mg per day, the next four days.
  Additional intramuscular injection of the drug Dalargin (solution for intravenous and intramuscular doses) under dosage of 1 mg daily once per day for 10 days
  Arms: group 2
Procedure: Standard therapy recommended by the Ministry of Health of the Russian Federation and Leitragin inhalation — Hydroxychloroquine + azithromycin + / - tocilizumab. Hydroxychloroquine intake is conducted according to the following schedule: 400 mg twice per day for 1-2 days of the treatment and 200 mg twice per day during six days of the treatment course.
  For the tocilizumab, 400 mg intravenously drip slowly (for at least 1 hour), with insufficient effect, administration is repeated the after 12 hours. Simultaneously no more than 800 mg of tocilizumab could be administered.
  For the azithromycin admission 500mg on day 1 is prescribed followed by 250mg per day, the next four days.
  Additional inhalation of the drug Leitragin, at a dose of 10 mg daily once per day until the symptoms of pulmonary complications will be ceased.
  Arms: group 3
Procedure: Standard therapy recommended by the Ministry of Health of the Russian Federation and Leitragin intramuscular injection combined with Leitragin inhalation — Hydroxychloroquine + azithromycin + / - tocilizumab. Hydroxychloroquine intake is conducted according to the following schedule: 400 mg twice per day for 1-2 days of the treatment and 200 mg twice per day during six days of the treatment course.
  For the tocilizumab, 400 mg intravenously drip slowly (for at least 1 hour), with insufficient effect, administration is repeated the after 12 hours. Simultaneously no more than 800 mg of tocilizumab could be administered.
  For the azithromycin admission 500mg on day 1 is prescribed followed by 250mg per day, the next four days.
  Additional inhalation of the drug Leitragin, at a dose of 10 mg daily once per day until the symptoms of pulmonary complications will be ceased.
  Additional intramuscular injection of the drug Dalargin (solution for intravenous and intramuscular doses) under dosage of 1 mg daily once per day for 10 days
  Arms: group 4

SUMMARY:
The purpose of the study is to evaluate an effectiveness of the drug Dalargin in combination with Leitragin for the prevention and treatment of severe pulmonary complications symptoms associated with severe and critical coronavirus infection cases (SARS COVID19, expanded as Severe acute respiratory syndrome Cоrona Virus Disease 2019 ).

Test drugs that will be administered to patients are:

* Leitragin, solution for inhalation administration,
* Dalargin, solution for intravenous and intramuscular administration.

DETAILED DESCRIPTION:
Research objectives are:

1. To study the effectiveness of the drug Leitragin, a solution for inhalation, for the prevention of severe pulmonary complications in patients with coronavirus infection (SARS-COVID-19);
2. To study the effectiveness of the drug Leitragin, a solution for inhalation, for the treatment of severe pulmonary complications in patients with coronavirus infection (SARS-COVID-19);
3. To study the effectiveness of the drug Dalargin, a solution for intravenous and intramuscular administration, for the prevention of severe pulmonary complications in patients with coronavirus infection (SARS-COVID-19);
4. To study the effectiveness of the drug Dalargin, a solution for intravenous and intramuscular administration, for the treatment of severe pulmonary complications in patients with coronavirus infection (SARS-COVID-19);
5. To evaluate the safety and tolerability of the use of the drug Leitragin, a solution for inhalation administration, for the prevention of severe pulmonary complications in patients with coronavirus infection (SARS-COVID-19);
6. To evaluate the safety and tolerability of the use of the drug Leitragin, a solution for inhalation administration, for the treatment of severe pulmonary complications in patients with coronavirus infection (SARS-COVID-19);
7. To evaluate the safety and tolerability of the use of the drug Dalargin, a solution for intravenous and intramuscular administration, for the prevention of severe pulmonary complications in patients with coronavirus infection (SARS-COVID-19);
8. To evaluate the safety and tolerability of the use of the drug Dalargin, a solution for intravenous and intramuscular administration, for the treatment of severe pulmonary complications in patients with coronavirus infection (SARS-COVID-19).

Upon admission to a specialized hospital for all patients with suspected COVID-19 Polymerase chain reaction (PCR) is being conducted. Only patients with confirmed coronavirus infection are included in the study.

It is an open, randomized clinical trial of the drug Dalargin in combination with Leitragin for the prevention and treatment of severe pulmonary complications symptoms in patients with coronavirus infection (SARS-COVID-19)

ELIGIBILITY:
Inclusion Criteria:

* Patients from the age of 18 years male and female;
* Coronavirus infection confirmed by results of Polymerase chain reaction test;
* Hospitalization of the patient;
* The presence of a signed informed consent to participate in the study.

Exclusion Criteria:

1. Revocation of informed consent by the patient.
2. Patient mismatch inclusion criteria.
3. First identified conditions and / or diseases described in the non-inclusion criteria.

The criteria for early termination of patient participation in the study during the period of use of the study drug are:

1. Patient withdrawal of informed consent.
2. First identified conditions and / or diseases described in the non-inclusion criteria.
3. The occurrence of serious adverse events.
4. Adverse events that do not meet the criteria of severity, the development of which, according to the researcher, further participation in the study may be detrimental to the health or well-being of the patient.
5. Administrative reasons (termination of the study by the Sponsor or regulatory authorities), as well as gross protocol violations that may affect the results of the study.
6. The patient receives / needs additional treatment that may affect the outcome of the study or patient safety
7. Individual intolerance to research drugs
8. Incorrect inclusion (for example, the patient was included in violation of the criteria for inclusion / non-inclusion of the protocol)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
The change of viral load in patients with SARS-COVID-19. | Upon patient inclusion in the study, after 96 hours and on the 10day;
  Estimated by Polymerase chain reaction (PCR)
The frequency of development of Acute Respiratory Distress Syndrome (ADRS) | up to 10 days
  Assessed through the entire patient participation in the study
Duration of hospitalization | up to 10 days
  The number of days a patient is hospitalized
The frequency of early mortality | up to 30 days
  Early mortality from all causes will be estimated
The frequency of late mortality | up to 90 days
  Late mortality from all causes will be estimated
Clinical status at the time of completion of participation in the study | an average of 10 days
  Clinical status at the time of completion of participation in the study will be estimated based upon the following criteria:
  1. Death;
  2. Hospitalization is extended, on invasive mechanical ventilation of the lungs with extracorporeal membrane oxygenation;
  3. Hospitalization extended, on non-invasive ventilation;
  4. Hospitalization is extended, needs additional oxygen;
  5. Hospitalization is extended, additional oxygen is not required;
  6. Discharged.

CONTACTS AND LOCATIONS:
Locations (1):
- Burnasyan Federal Medical Biophysical Center FMBA of Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No